CLINICAL TRIAL: NCT07237568
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy and Safety of LNK01001 in Adult Subjects With Active Ankylosing Spondylitis
Brief Title: A Study to Evaluate Efficacy and Safety of LNK01001 in Adults With Ankylosing Spondylitis
Acronym: AS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lynk Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LK001302
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Ankylosing Spondylitis
Keywords: LNK01001; AS
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LNK01001 12mg (Experimental): Participants receive LNK01001 12mg orally BID for 52 weeks.
  Interventions: Drug: LNK01001
- Placebo (Placebo Comparator): Participants receive matching placebo for 16 weeks and then switch to receive LNK01001 12mg orally BID for 36 weeks.
  Interventions: Drug: LNK01001; Drug: Placebo

INTERVENTIONS:
Drug: LNK01001 — Capsule; Oral
Drug: Placebo — Capsule; Oral
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of LNK01001 in subjects with active ankylosing spondylitis.

The study is comprised of a 16-week randomized, double-blind, parallel-group, placebo-controlled period (the Double-Blind Period); a 36-week open-label, long-term extension period (the Open-Label Extension Period). In the Double-Blind Period, participants will be randomized in a 1:1 ratio to receive either LNK01001 or placebo twice daily (BID). Participants in the placebo group will be switched to LNK01001 BID at Week 16 in the Open-Label Extension Period.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of ankylosing spondylitis (AS) and meet the modified New York Criteria for AS.
* Participant must have a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥ 4 at the Screening and Baseline Visits and Must have a Total Back Pain score ≥ 4 based on a 0 - 10 numerical rating scale at the Screening and Baseline Visits.
* Has had an inadequate response to at least 2 nonsteroidal anti-inflammatory drugs (NSAIDs) over an at least 4-week period in total at maximum recommended or tolerated doses, or has an intolerance to or contraindication for NSAIDs as defined by the Investigator.

Exclusion Criteria:

* Total spinal ankylosis.
* Participants with known allergies to components or excipients of the study drug.
* Requirement of prohibited medications during the study.
* Participants who are pregnant, nursing, or planning a pregnancy during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Assessment of SpondyloArthritis International Society 40 (ASAS40) Response at Week 16 | Baseline and week 16
  ASAS40 response was defined as improvement of ≥ 40% relative to Baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a net worsening of > 0 units) in the potential remaining domain:
  * Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain);
  * Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).

SECONDARY OUTCOMES:
Percentage of Participants Achieving Assessment of SpondyloArthritis International Society 20 (ASAS20) Response at Week 16 | Baseline and week 16
  ASAS20 response was defined as an improvement of ≥ 20% and an absolute improvement of ≥ 1 unit (on a scale of 0 to 10) from Baseline in at least 3 of the following 4 domains, with no deterioration (defined as a worsening of ≥ 20% and a net worsening of ≥ 1 units [on a scale of 0 to 10]) in the remaining domain:
  * Patient's global assessment of disease activity, measured on a NRS from 0 (no activity) to 10 (severe activity);
  * Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain);
  * Function, measured by the BASFI which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible);
  * Inflammation, measured by the mean of the 2 morning stiffness-related BASDAI NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Percentage of Participants With Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response at Week 16 | Baseline and week 16
  The BASDAI assesses disease activity by asking the participant to answer 6 questions (each on an 11 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For Questions 1 to 5 (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
  A BASDAI 50 response is defined as improvement of 50% or more from Baseline in BASDAI score.
Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 16 | Baseline and week 16
  ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  1. Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe])
  2. Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity])
  3. Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe])
  4. Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours])
  5. High-sensitivity C-reactive protein (hs-CRP) in mg/L. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS include Inactive disease (ASDAS < 1.3) and very high disease (ASDAS > 3.5). A negative change from Baseline score indicates improvement in disease activity.
Percentage of Participants With ASDAS Inactive Disease at Week 16 | Baseline and week 16
  ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  1. Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe])
  2. Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity])
  3. Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe])
  4. Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours])
  5. High-sensitivity C-reactive protein (hs-CRP) in mg/L. The overall score ranges from 0 with no defined upper score. ASDAS Inactive Disease is defined as an ASDAS score < 1.3.
Change From Baseline in Patient's Assessment of Total Back Pain at Week 16 | Baseline and week 16
  Participants assessed their total back pain during the last week on a 0 to 10 numerical rating scale (NRS), where 0 represents no pain and 10 represents most severe pain.
Change From Baseline in Patient's Assessment of Nocturnal Back Pain at Week 16 | Baseline and week 16
  Participants assessed the amount of back pain at night over the last week on a 0 to 10 NRS, where 0 represents no pain and 10 represents most severe pain.
Percentage of Participants With ASDAS Low Disease Activity at Week 16 | Baseline and week 16
  ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  1. Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe])
  2. Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity])
  3. Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe])
  4. Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours])
  5. High-sensitivity C-reactive protein (hs-CRP) in mg/L. The overall score ranges from 0 with no defined upper score. ASDAS Low Disease Activity is defined as an ASDAS score < 2.1.
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 16 | Baseline and week 16
  The Bath Ankylosing Spondylitis Functional Index is a validated index to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities such as putting on socks, bending, reaching, getting up from the floor or an armless chair, standing, climbing and other physical activities. Each item is scored on a NRS ranging from 0 (easy to perform an activity) to 10 (impossible to perform an activity). The overall score is the mean of the 10 items and ranges from 0 to 10 with higher scores indicating more functional limitations. A negative change from Baseline in BASFI indicates improvement.
Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Score at Week 16 | Baseline and week 16
  The ASQoL consists of 18 items related to quality of life, including the impact of pain on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. Each item is answered as yes (scored as 1) or no (scored as 0).
  Scores are summed to obtain the overall score which ranges from 0 to 18, where higher scores indicate a worse quality of life. A negative change from Baseline in ASQoL indicates improvement in quality of life.
Change From Baseline in Linear Bath Ankylosing Spondylitis Metrology Index (BASMI) at Week 16 | Baseline and week 16
  The BASMI is a composite score based on 5 direct measurements of spinal mobility:
  1. cervical rotation (measured in degrees),
  2. tragus to wall distance (in centimeters [cm])
  3. lumbar side flexion (in cm),
  4. lumbar flexion (modified Schober's) (in cm) and
  5. intermalleolar distance (in cm). Each measurement is converted to a linear score between 0 and 10. The total BASMI score is the average of the 5 scores and ranges from 0 to 10; the higher the BASMI score the more severe the patient's limitation of movement due to their ankylosing spondylitis. A negative change from Baseline indicates improvement.
Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 16 | Baseline and week 16
  The MASES evaluation was conducted to assess the presence or absence of enthesitis (inflammation of the entheses, or sites where tendons or ligaments insert into the bone) at 13 different sites (first costochondral joint left/right, seventh costochondral joint left/right, posterior superior iliac spine left/right, anterior superior iliac spine left/right, iliac crest left/right, fifth lumbar spinous process, and proximal insertion of Achilles tendon left/right. Each site was scored for presence (1) or absence (0) of enthesitis. The MASES is the sum of the 13 site scores, and ranges from 0 to 13, with higher scores indicating more inflammation of the entheses. A negative change from Baseline indicates improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No